CLINICAL TRIAL: NCT05369923
Title: Survey of Knowledge and Attitude of Pain in Anesthesia Residents of Thailand
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: REC.65-038-8-1
Record Dates: First submitted 2022-04-21; First posted 2022-05-11 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective descriptive cross-sectional survey using the modified Knowledge and Attitudes Survey Regarding Pain (KASRP) in English via an online google form.

DETAILED DESCRIPTION:
Setting of the study/Trial site This study will be conducted via google form survey.

Target population (Provide a complete description of your target population in the study) Anesthesia residents of all levels throughout Thailand.

Study population (Provide details of your population in the study) Anesthesia residents of all levels throughout Thailand.

Inclusion criteria Anesthesia residents of all levels throughout Thailand.

Exclusion criteria Anesthesia residents who do not want to participate in this study.

Withdrawal criteria (e.g. research participant withdrawal, adverse outcome during participating the study) Anesthesia residents can stop answering the questionnaire survey at any time.

Termination criteria (e.g. terminating investigational product treatment/trial treatment) Not relevant

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residents of all levels throughout Thailand.

Exclusion Criteria:

* Anesthesia residents who do not want to participate in this study.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anesthesia residents in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain knowledge | Through study completion, an average of 1 year
  To measure knowledge of pain management by using the "Knowledge and Attitudes Survey Regarding Pain" (KASRP) questionnaire which consists of 39 questions (the higher number of correct answers, the better)

SECONDARY OUTCOMES:
Pain attitude | Through study completion, an average of 1 year
  To measure attitudes of pain management by using the "Knowledge and Attitudes Survey Regarding Pain" (KASRP) questionnaire which consists of 39 questions (the higher number of correct answers, the better)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim MH, Park H, Park EC, Park K. Attitude and knowledge of physicians about cancer pain management: young doctors of South Korea in their early career. Jpn J Clin Oncol. 2011 Jun;41(6):783-91. doi: 10.1093/jjco/hyr043. Epub 2011 Apr 18. PMID 21502282